CLINICAL TRIAL: NCT06893146
Title: Protocol for a Quasi-experimental Controlled Study to Reduce Sedentary Lifestyle in Patients With Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of La Rioja (Other)
Responsible Party: Principal Investigator, Raquel Sainz Prado, Principal Investigator, University of La Rioja
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI 778
Record Dates: First submitted 2025-03-11; First posted 2025-03-25 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Sedentary Behaviors
Keywords: Diabetes; Sedentary lifestyle; Sedentary behavior; quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sedentary Behavior; Diabetes Mellitus | interventions — Training Support

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This group will receive face-to-face group and individual visits and telephone calls.
  Interventions: Behavioral: Reduction of Sedentary Behavior
- Control group (Active Comparator): The control grup will receive every two months written information on healthy lifestyle habits by e-mail.
  Interventions: Behavioral: Educational support

INTERVENTIONS:
Behavioral: Reduction of Sedentary Behavior — The intervention group will receive an intervention that will include two group sessions, bimonthly phone calls and a face-to-face visit with the study nurse. Phone calls will be made every two months using motivational interviewing techniques with the aim of educating on habits and behaviors that reduce sedentary lifestyles, addressing needs and concerns on an individual basis, and enhancing patients motivation, well-being and quality of life. The same purpose is served by the face-to-face visit that will be conducted in the third month of the study. The study's interventions have a personalized approach, which considers individual preferences and needs to consolidate the new habits acquired in the long term. The active intervention has a duration of 6 months and will be carried out by nursing professionals.
  Arms: Intervention group
Behavioral: Educational support — Every two months, this group will receive detailed written information about healthy lifestyle habits via email, emphasizing the importance of maintaining an active lifestyle. Additionally, they will be provided with standard educational material on the management of type 2 diabetes.
  Arms: Control group

SUMMARY:
The prevalence of diabetes has increased worldwide, making it the most prevalent metabolic disorder. Physical inactivity contributes to the progression of this disease and aggravates other comorbidities, such as obesity and cardiovascular disease. Beneficial strategies aimed at promotion and healthy aging, oriented to decrease sedentary behavior, are necessary to obtain desirable metabolic effects and improve the quality of life of people with diabetes.

The objective is to examine, through a clinical trial, the effect of decreasing sedentary time and increasing motivation to adopt an active lifestyle on different clinical, anthropometric and biochemical parameters in patients diagnosed with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
A quasy-experimental controlled study with a 12-month follow-up will be carried out. The study has been chosen to be conducted as a single-center study for strategic and logistical reasons. A two-arm parallel design will be used. The control group (CG) will receive messages by mail with healthy lifestyle habits, while the intervention group (IG) will receive a behavioral intervention based on lifestyle modification, focusing on reducing sedentary time. These interventions will be directed by the research nurse.

The general objective of the study is to know the effect of decreasing sedentary time and increasing motivation to adopt an active lifestyle of different health-related parameters in patients diagnosed with type 2 diabetes mellitus. Also to provide support and resources for the proper management of diabetes. Likewise, it will be verified that face-to-face interventions and telephone interventions by nursing professionals decrease the sedentary time in the diabetic population and if it means and improvement in clinical, anthropometric and biochemical parameters. Also, to evaluate the quality of life and the degree of motivation aimed at reducing sedentary time and to integrate the reduction of sedentary time in the lifestyle of the participants with practical tools and guidelines adapted to the circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus
* 18 years of age or older
* Minimal physical fitness

Exclusion Criteria:

* Medical contraindication
* Pregnant women
* Recent surgical interventions limiting mobility
* Patients currently undergoing oncological treatment or less than one year since the end of treatment.
* Suffering from dementia, impairment or a severe cognitive or psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Level of sedentary lifestyle | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  The level of sedentary lifestyle will be measured with the use of accelerometers.
  The model used in our study is ActiTrainer.
Level of sedentary lifestyle | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  The level of sedentary lifestyle will be measured with the questionnaire validated in Spanish Sedentary Behavior Questionnaire. This instrument measures the time spent on sedentary behaviors from the moment the person wakes up until they go to bed, performed during weekdays and weekends. Responses are provided on numerical scales, and then the total number of hours dedicated to each activity is summed up. Higher scores indicate more time spent in sedentary activities.
State of motivation to change | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Measured by the Transtheoretical Model of Physical Exercise Change Questionnaire. This questionnaire identifies the stage of the Transtheoretical Model of Change in which a person stands regarding their willingness to engage in physical exercise. It consists of two tables: one for those who do not exercise regularly, with items about reasons for not exercising, and another for those who do, with reasons for exercising. Responses are rated on a scale from 1 (strongly disagree) to 5 (strongly agree). The measurement is based on the average scores for each stage of the model. Higher scores indicate a greater readiness to engage in physical activity (better outcome in terms of behavior change).

SECONDARY OUTCOMES:
Physical activity level | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  To measure the level of physical activity, the short, self-administered format of the "International Physical Activity Questionnaire" will be used.
  Questions are asked about the time spent on activity over the past 7 days, distinguishing between vigorous activities, walking, or sitting. Results are calculated in minutes per week by multiplying the number of days by the duration of the activity in minutes, obtaining a weekly value for each category. A person is considered inactive if they do not meet the recommended threshold of 150 minutes of moderate physical activity per week. They are classified as sufficiently active if they reach 150 minutes of moderate or 75 minutes of vigorous activity per week, and very active if they exceed 300 minutes of moderate or 150 minutes of vigorous activity per week, as recommended by the WHO.
Quality of life in people with diabetes | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  The validated Spanish version of the Diabetes Quality of Life Questionnaire (DQoL) will be used. Participants rate the items on a 5-point Likert scale, where 1 represents "strongly disagree" and 5 represents "strongly agree." Other items are rated from 1 ("very satisfied") to 5 ("very dissatisfied"). The scores are quantified, with higher scores indicating better quality of life, while lower scores suggest a greater negative impact of diabetes on the patient's life.

OTHER OUTCOMES:
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Levels of glucose: mg/dL (milligrams per deciliter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Glycosylated hemoglobin (HbA1c): % (percentage).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Homeostasis model assessment-insulin resistance (HOMA-IR): Dimensionless unit.
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Total cholesterol: mg/dL (milligrams per deciliter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  High-density lipoprotein cholesterol (HDL-c): mg/dL (milligrams per deciliter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Low-density lipoprotein cholesterol (LDL-c): mg/dL (milligrams per deciliter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Triglycerides (TG): mg/dL (milligrams per deciliter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Aspartate aminotransferase (AST): U/L (units per liter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Alanine aminotransferase (ALT): U/L (units per liter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Gamma-glutamyl transferase (GGT): U/L (units per liter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Creatinine: mg/dL (milligrams per deciliter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Urea: mg/dL (milligrams per deciliter.
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Creatinine clearance: mL/min (milliliters per minute).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Iron: µg/dL (micrograms per deciliter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Ferritin: ng/mL (nanograms per milliliter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Sodium: mmol/L (millimoles per liter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Potassium: mmol/L (millimoles per liter).
Clinical characteristics | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  C-reactive protein (CRP): mg/L (milligrams per liter).
Blood pressure | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Measurements will be taken over the brachial artery, after 5 minutes of rest while seated and with the arms resting at heart level. Long-sleeved shirts will be removed for a correct reading and the cuff size must be adequate.
Anthropometric data | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Anthropometric measurements of weight are collected by healthcare personnel using calibrated instruments and clinical standard procedures. Weight will be measured in kilograms (kg).
Anthropometric data | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Anthropometric measurements of height are collected by healthcare personnel using calibrated instruments and clinical standard procedures. Height will be measured in centimeters (cm).
Anthropometric data | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Weight and height will be combined to report the BMI in kg/m².
Anthropometric data | At baseline, and at 3, 6 and 12 months after the initiation of the intervention
  Anthropometric measurements of waist-hip circumference are collected by healthcare personnel using calibrated instruments and clinical standard procedures. Waist-hip circumference will be measured in centimeters (cm).

REFERENCES:
- [Derived] Sainz-Prado R, Sainz-Prado A, Andrade-Gomez E, Rodriguez-Roca B. Quasi-experimental controlled study protocol to reduce sedentary lifestyle in patients with type 2 diabetes. PLoS One. 2025 Sep 16;20(9):e0330393. doi: 10.1371/journal.pone.0330393. eCollection 2025. PMID 40956797